CLINICAL TRIAL: NCT01157390
Title: Tolerance and Efficacy of Wondersun Infant Formula in Formula-fed Chinese Term Infants: an Open Label, Controlled Trial
Brief Title: Tolerance and Efficacy of Wondersun Infant Formula in Formula-fed Chinese Term Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Enzymotec (Industry)
Responsible Party: Principal Investigator, Yu-ming Chen, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INF-004
Record Dates: First submitted 2010-06-24; First posted 2010-07-07 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Infant Nutrition
Keywords: Term-infant; sn-2 palmitic acid; infant formula
MeSH Terms: interventions — Infant Formula; Lactation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infant formula (Experimental): The infants will be fed with Wondersun infant formula with high proportion of palmitic acid at the sn-2 position
  Interventions: Other: Infant formula
- Breast feeding (Active Comparator): Complete breast feed within the first 3 month
  Interventions: Other: Breast feeding

INTERVENTIONS:
Other: Infant formula — Name: Infant formula with high proportion of palmitic acid in the sn-2 position Dosage & frequency: Fed as need Duration: at least 3 months
  Other Names: Wondersun Brand An Li Cong Infant Formula
  Arms: Infant formula
Other: Breast feeding — Breast feeding
  Other Names: Not relevant
  Arms: Breast feeding

SUMMARY:
Objective: To demonstrate the well-being of Chinese term infants fed with Wondersun formula with high proportion of palmitic acid in the sn-2 position.

Design & setting: A single-center, open label study. A breast fed group will serve as reference. The study will be conducted in Guangzhou from 2010.1~2010.12.

Participants: 0-14 d whole formula-fed infants and whole breast-fed infants, 30 infants in each group. They are required to be healthy, term-infant, and with normal birth weight, and have no medications known to affect their growth and development.

Intervention: The formula-fed infants will be fed Wondersun formula with high proportion of palmitic acid in the sn-2 position; and breast-fed groups will be fed using breast milk for at least 3 month.

Outcome measures: Tolerance and efficacy will be assessed by body measurement, stool characteristics questionnaire, general health examination, and behavior and habit questionnaire at baseline (0-14d), 6 weeks and 12 weeks. Safety will also be evaluated.

Statistical analysis: t-test, rank test and chi-square test will be used to examine the significance of change from baseline to follow-up visit between the formula-fed and breast-fed groups for effectiveness measures

ELIGIBILITY:
Inclusion Criteria:

* Parental/legal guardian written informed consent.
* The mother had unequivocally decided not to breast-feed (for formula fed infants) or to breastfeed (for human milk fed infants).
* Term infant of Chinese origin born at 37-42 gestation weeks as determined by menstrual history and corroborated by prenatal Unltra-Sound (US) and/or physical examination.
* Birth weight appropriate for gestational age (AGA), 2500-4000g (between 10th~ 90th percentile of body weight at same gestation age).
* The infant is apparent healthy at birth and entry to study.
* Apgar after 5 minutes >7.
* Enrolled within their first 14 days after birth.
* The infant is a product of normal pregnancy and delivery including C-section.
* Patental ability to attend visits, interviews and willing to fill questionnaires.

Exclusion Criteria:

* Mother health condition: (psychological of physical) or socioeconomic problems that may interfere with the mother's ability to take care of her infant.
* The infant suffers from a major congenital abnormality or chromosomal disorder with a clinical significance that can be detected at birth.
* The infant suffers/ed from a disease requiring mechanical ventilation or medication treatment at the first week after birth.
* The infant suffers from any suspected or known metabolic or physical limitations interfering with feeding or normal metabolism (require a special formula).
* The infant is a carry of HBV (HBsAb positive).

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Anthropometric parameters | 12 weeks
  body length, body weight, and head circumferences

SECONDARY OUTCOMES:
Efficacy and safety | 6 weeks
  Stool characteristics General health and wellbeing Behavior and habits Adverse events Concomitant medications Covariates or potential confounders

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Chen, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Zhong W, Tang XY, Hou HY, Liora L, Yael L, Yonatan M, Fabiana BY, Wei M, Su YX, Chen YM.Tolerance and Efficacy of Infant Formula with High Sn-2 Palmitate in Formula- Fed Chinese Term Infants: an Open Label, Controlled Trial. J Nutr Health Food Eng 2016 Mar 15; 4(2): 00122. DOI: 10.15406/jnhfe.2016.04.00122